CLINICAL TRIAL: NCT05157906
Title: Effects of the Happy Grow Program on Parental Self-confidence: A Randomized, Controlled Open-label Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20.29.INF
Record Dates: First submitted 2021-10-07; First posted 2021-12-15 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Responsive Parenting

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled education-based interventional study without any investigational product. Study subjects are randomized to the intervention or control groups with a follow-up period of 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Subjects will have access to the Grow Happy program materials, including the Grow Happy Book, 99+ Ways to Grow Happy Tips and Engagement Videos, which are provided digitally during the trial duration of 12 weeks.
  Interventions: Behavioral: Education based
- Control Group (Active Comparator): No additional education materials will be proactively provided during trial duration. Subjects will only be provided with the Indonesian standard of care only.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Education based — The interventional materials will be provided digitally for 12 weeks, with the monthly theme featured from the educational Grow Happy book and related tips and videos that will be released weekly.
  Arms: Experimental Group
Behavioral: Control — At enrollment, subject will be provided with the Mother and Child booklet, which is the Indonesian standard of care for parenting guidance.
  Arms: Control Group

SUMMARY:
This is a randomized, controlled education-based interventional study without any investigational product. Study subjects are randomized to the intervention or control groups with a follow-up period of 12 weeks. 250 toddlers between ages 24 and 28 months with first-time primary caregiver (mother or father) from low to mid-income families in Indonesia will be enrolled.

DETAILED DESCRIPTION:
Extensive scientific literature demonstrates that childhood happiness can be nurtured through positive and responsive parenting strategies, and is associated with optimal child development and is a predictor of future happiness.

The Grow Happy program is a translation of scientific literature into parent-friendly educational materials and actionable tips and advice aimed at improving parental knowledge and child happiness through parenting techniques and play.

Although the Grow Happy Program is scientifically validated, it has yet to be clinically tested. It is hypothesized that the Grow Happy program will improve mothers' knowledge and self-confidence related to parenting behaviors that promote happiness and optimal child development.

ELIGIBILITY:
Inclusion criteria:

1. Caregiver-toddler dyad pair is from low to mid-income households, as defined by a cut-off annual income level of IDR <4,800,000 according to National Socioeconomic Survey.
2. Toddlers (full-term) between ages of 24 and 28 months at time of enrolment.
3. Normally developing toddlers without any diagnosed behavioral, neurological or eating issues.

Exclusion criteria:

1. Primary caregivers with more than one child.
2. Primary caregivers with diagnosed behavioral or eating issues.
3. Toddlers with weight-for-age value < -2 SD from the National Indonesian Growth Chart or per WHO Standards at enrollment.
4. Toddlers with height-for-age < -2 SD from the National Indonesian Growth Chart or per WHO Standards at enrollment.

Ages: 24 Months to 28 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
To increase self-confidence of mothers (vs. control group) to adopt responsive parenting behaviors that promote optimal child development. | Change from baseline (V1) to 12 weeks of intervention (V2).
  Mothers' self-confidence based on composite scores from the Toddler Care Questionnaire.

SECONDARY OUTCOMES:
Parenting experience | Change from baseline to 12 weeks
  Parenting Experience Questionnaire based on composite scores from a self-administered Questionnaire.
Child's health-related quality of life | Change from baseline to 12 weeks
  Child's health related quality of life scores from the Infant and Toddler Quality of Life Questionnaire Short Form (ITQOL-SF47).
Maternal health-related quality of life | Change from baseline to 12 weeks
  Maternal health related quality of life scores from the Oxford Happiness Inventory (OHI).
Toddler gut comfort | Change from baseline to 12 weeks
  GI symptoms, behaviors and overall GI burden assessed using the Toddler Gut Comfort Questionnaire.
Child eating behavior | Change from baseline to 12 weeks
  Child eating behaviors and patterns assessed using the Child-Parent Mealtime Behavior Questionnaire.
Child temperament | Change from baseline to 12 weeks
  Child temperament as assessed by Children's Behavior Questionnaire (CBQ) Short Form.
Child playfulness | Change from baseline to 12 weeks
  Child playfulness as measured by the Playfulness Questionnaire.
Parenting responsiveness behaviors | Change from baseline to 12 weeks
  Parenting responsiveness using the parenting scale derived from the Parenting Young Children Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Juffrie Mohammad, Ph.D., SpAK, Principal Investigator — Faculty of Medicine, Public Health and Medicine, Universitas Gadjah Mada
Locations (1):
- University Gadjah Mada, Center for Health and Human Nutrition, Sleman, Indonesia